CLINICAL TRIAL: NCT00249041
Title: Open-label Study to Assess the Antibody Response to Etanercept Liquid in Subjects With Rheumatoid Arthritis (RA)
Brief Title: Enbrel Liquid Immunogenicity Protocol
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Immunex Corporation (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20050145
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Last update posted 2010-07-30 (Estimated); Status verified 2010-07

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis, Enbrel liquid, antibodies
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept

ARMS (1):
- Etanercept liquid (Experimental)
  Interventions: Drug: 50 mg Etanercept; Drug: Enbrel liquid

INTERVENTIONS:
Drug: 50 mg Etanercept — 50 mg Etanercept liquid injected SC once weekly using prefilled syringes
Drug: Enbrel liquid — 50 mg Etanercept liquid injected SC once weekly using prefilled syringes

SUMMARY:
The purpose of this study is to assess the antibody formation to Enbrel liquid in subjects with Rheumatoid Arthritis

DETAILED DESCRIPTION:
The purpose of this study is to assess the rate of anti-etanercept antibody formation in a larger sample of subjects on liquid etanercept than the previous study, 20020378, in a minimum of 400 subjects receiving etanercept liquid for the first time, with and without concomitant MTX therapy. The rate of neutralizing antibodies to liquid etanercept will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Must be able to self-inject or have someone who can do so for them
* Should have Rheumatoid Arthritis per ARA criteria and screening lab results per predefined value

Exclusion Criteria:

* Any prior biologic therapy for inflammatory disease
* Any prior cyclophosphamide therapy
* Not using adequate contraception
* Pregnant or breast-feeding or any significant concurrent medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 447 (Actual)
Dates: Start 2005-10; Primary Completion 2006-12 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Rates of anti-etanercept antibody formation to etanercept liquid with or without concomitant methotrexate (MTX) therapy at week 24 | 24 weeks

SECONDARY OUTCOMES:
Rates of anti-etanercept antibody formation to etanercept liquid at week 12, and the rates of neutralizing antibodies at Weeks 12 and 24. Safety of etanercept liquid in RA subjects receiving 50 mg once weekly up to 24 weeks. | 12 weeks and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Kavanaugh A, Lee SJ, Weng HH, Chon Y, Huang XY, Lin SL. Patient-derived joint counts are a potential alternative for determining Disease Activity Score. J Rheumatol. 2010 May;37(5):1035-41. doi: 10.3899/jrheum.090704. Epub 2010 Feb 15. PMID 20156946
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_916_ENBREL_20050145.pdf
- See also: FDA-approved Drug Labeling — http://www.enbrel.com/
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com